CLINICAL TRIAL: NCT03471741
Title: Moderated Accelerated RAdiotherapy (MARA-2) in Moderate-high Risk Breast Cancer: a Phase I-II Study
Brief Title: Intensity Modulated Radiotherapy With Concomitant Boost in Breast Cancer
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: MARA-2
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer; Radiation Toxicity
Keywords: breast cancer; radiotherapy; cutaneous toxicity; subcutaneous toxicity; local control; IMRT
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MARA-2: IMRT with concomitant boost: A forward planned IMRT technique was used and the prescribed dose to the whole breast was 50 Gy plus a concomitant boost of 10 Gy to the tumor bed
  Interventions: Radiation: IMRT with concomitant boost
- CG: 3D-RT with sequential boost: The whole breast received 50.4 Gy in 28 fractions delivered with 3D-RT, followed by a sequential boost on the tumor bed of 10 Gy in 4 fractions delivered with electrons
  Interventions: Radiation: 3D-RT with sequential boost

INTERVENTIONS:
Radiation: IMRT with concomitant boost
  Groups: MARA-2: IMRT with concomitant boost
Radiation: 3D-RT with sequential boost
  Groups: CG: 3D-RT with sequential boost

SUMMARY:
To assess feasibility of postoperative IMRT with concomitant boost in moderate-high risk breast cancer in terms of late toxicity and local control

DETAILED DESCRIPTION:
Patients treated conservatively with moderate-high risk breast cancer were treated with IMRT plus concomitant boost to surgical bed (up to a dose of 50 Gy to whole breast and 60 Gy to the tumor bed).

Aim of the study was to evaluate late toxicity and local control after this treatment compared with a historical control group (CG) of patients treated with 3D-conformal postoperative radiotherapy delivered with conventional fractionation.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed invasive breast cancer (pT1-4) with at least one of these characteristics: 3 or more metastatic axillary nodes, pre or peri-menopausal status, close resection margins
* breast conservative surgery

Exclusion Criteria:

* positive margins
* distant metastases

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From 2003, all women fullfilling the inclusion criteria were treated with MARA-2 scheme
Sampling Method: Non-Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2001-06-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment.related late adverse events | 5 years
  late toxicity (cutaneous and subcutaneous) is evaluated using RTOG/EORTC criteria in both groups of patients

SECONDARY OUTCOMES:
Local control | 5 years
  absence of locoregional relapse

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G Morganti, MD, Principal Investigator — Radiation Oncology Center, Department of Experimental, Diagnostic and Speciality Medicine-DIMES, Unversity of Bologna, S. Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Macchia G, Cilla S, Buwenge M, Zamagni A, Ammendolia I, Zamagni C, Frezza GP, Valentini V, Deodato F, Morganti AG. Intensity-Modulated Radiotherapy with Concomitant Boost After Breast Conserving Surgery: A Phase I-II Trial. Breast Cancer (Dove Med Press). 2020 Nov 12;12:243-249. doi: 10.2147/BCTT.S261587. eCollection 2020. PMID 33209058